CLINICAL TRIAL: NCT05818202
Title: Experiences, Attitudes, and Perspectives of Stroke Patients and Physiotherapists in Robotic Rehabilitation
Brief Title: Perspections of Stroke Patients and Physiotherapists in Robotic Rehabilitation
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Güzin Kara, PT. PhD. Assist. Prof., Pamukkale University
Other Study IDs: E-60116787-020-113947
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Paralysis; Physician's Role
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: The stroke patients who can understand the questionnaires, have only a stroke history, and not have another neurological condition which affect the study.
  Interventions: Other: Questionannire
- Physiotherapists: Physiotherapists graduated from a university with at least a bachelor degree of physiotherapy and rehabilitation and work in Denizli.
  Interventions: Other: Questionannire

INTERVENTIONS:
Other: Questionannire — The questionannaires for both physiotherapists and stroke patients were formed in this study. The perspectives of the participants were recorded.

SUMMARY:
This study was a cross-sectional study. The insights of stroke patients and physiotherapists were assessed with the quantitative questionnaires. The results were provided as number, percentage, mean, and standard deviation. The results of the insights of the current sapmle were given and compared the previous studies. The authors though that the results of the study can fill the gaps in robotic rehabilitation and support a better robotic rehabilitation experience.

DETAILED DESCRIPTION:
Fifty stroke patients and fifty seven physiotherapists included the study. A seventeen-item and eight-item questionnaire s were created for stroke patients and physiotherapists, respectively. The descriptive data of the stroke patients and physiotherapists were presented. The results were compared with the literature and interpreted to guide future studies.

ELIGIBILITY:
For stroke patients

Inclusion Criteria:

* Having a single stroke

Exclusion Criteria:

* Having a communication problem
* Having another neurological condition which can affect the study

For physiotherapists

Inclusion Criteria:

* Graduating from a physiotherapy and rehabilitation program with at least a bachelor degree
* Working in Denizli

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty stroke patients and fifty seven physiotherapists were participated in the study. All participants met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
A seventeen-item questionnaire | 1 year
  The items of the questionnaires were depends on investigating of the perspectives, attitudes, and experiences of stroke patients.
An eight-item questionnaire | 1 year
  The items of the questionnaires were depends on investigating of the perspectives, attitudes, and experiences of physiotherapists.

CONTACTS AND LOCATIONS:
Overall Officials: Güzin Kara Çakıcı, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)